CLINICAL TRIAL: NCT03920345
Title: Endoscopic Electrothermic Procedure of the Sacroiliac Joint
Acronym: ESIJ
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participation.
Sponsor: joimax, Inc. (Industry)
Collaborators: MileStone Research Organization (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MULTI-2018-05-31
Record Dates: First submitted 2019-04-02; First posted 2019-04-18 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Chronic Lower Back Pain (CLBP); SIJ Arthropathy

STUDY DESIGN:
Intervention Model Description: A prospective, non-randomized, multi-center study, case series, clinical observation study of minimally invasive surgery for the treatment of SIJ arthropathy and chronic lower back pain (CLBP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment: Endoscopic ET on SI joint (Experimental): New techniques have been developed and tested to expand the usefulness of minimally invasive spine surgery beyond disk herniation. This includes endoscopic electrothermic ablation which can be used to target SIJ-associated CLBP. A small retrospective study demonstrated significant improvements in Visual Analog Scale and Oswestry Disability Index from pre-operative levels in patients with CLBP associated with the SIJ for up to 21 months following the procedure. However, there has not yet been a prospective study to assess the efficacy of this procedure, and therefore, this is the aim of this study.
  Interventions: Device: MultiZYTE

INTERVENTIONS:
Device: MultiZYTE — Subjects can be treated either unilateral or bilateral, depending on their condition and the recommended treatment by the surgeon. The decision is a clinical one and is not influenced by the decision of whether to be included in the study or the subsequent outcomes and QoL analysis.

SUMMARY:
1. Determine the rate and incidence of peri-operative & post-operative adverse events (complications, infections, re-operations, re-admissions) in the endoscopic approach for the treatment of SIJ arthropathy and chronic lower back pain (CLBP).
2. Determine the Health-Related Quality of Life (HRQoL) using EQ-5D scale, VAS (Visual Analog Scale) & ODI (Oswestry Disability Index), outcomes following the endoscopic approach for the treatment of SIJ arthropathy and chronic lower back pain (CLBP) (pre- to post-operative changes).

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) that lasts for more than six months is estimated to occur in 60-80% of the general population in their lifetime and is associated with substantial healthcare costs. The sacroiliac joint (SIJ) complex is one of the major sources of CLBP, accounting for around 10-33% of the total number of CLBP cases. The SIJ complex consists of the joint capsule, synovia, various muscles and ligamentous structures overlying the join and neuronal structures that innervate the SIJ. Current interventional and surgical treatment options for SIJ complex mediated CLBP include intraarticular and periarticular injection of the joint, SIJ fusion and radio frequency ablation (RFA) of the neuronal structures innervating the SIJ. The described interventional procedures are simple procedures and provides quick pain relief, but the effect is short-lived. In addition, SIJ fusion is an invasive surgical procedure that should be reserved for refractory intractable pain of the SIJ1.

New endoscopic electrothermic ablation of the SIJ capsula, synovial and neuronal structures have been utilized in the treatment of facetogenic CLBP in a few number of clinical reports with favorable results, but to our knowledge, the efficacy of this technique when applied to SIJ-associated CLBP has not been reported. In this study, the investigators will utilize endoscopy for the precise microsurgical and ablation (ESIJ) of the potential pain generators associated with the SIJ and evaluate the clinical efficacy of this new technique.

ELIGIBILITY:
Inclusion Criteria:

Subject age 18 - 85 years;

* SIJ arthropathy and chronic lower back pain (CLBP);
* Patient to undergo endoscopic electrothermic ablation of spinal levels S1-S3. The L4-L5 and/or L5-S1 facet joint can be included in the ablation per doctor discretion.
* Correct spinal levels (ranging L4-S3) to be treated have been confirmed by 1) diagnostic SIJ injection, followed by 2) diagnostic Medial/Lateral Branch Block at the applicable levels.
* The subject is likely to follow standard of care post-operative follow-up for at least 24 months.

Exclusion Criteria:

Patients receiving additional invasive back surgery after the study treatment.

* Inability to complete follow-up visits or required questionnaires.
* Non-compliant patients
* Difficult or impossible communication with the patient
* Breastfeeding, pregnant or patients who plan a pregnancy while participating in the study
* Systemic neurological disorders with mobility limitations (e.g. advanced Parkinson's disease or multiple sclerosis)
* Patients with incompatibilities or known limitations that make participation impossible
* Patients after stabilization with implants on thoracic or lumbar spine.
* Inability to provide informed consent without a legally authorized representative.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Change in EQ-5D-3L | Pre-Op, Peri-Op, 6-weeks, 3-months, 6-months, 12-months, 24-months post-op
  5 Question Health Questionnaire: patient's rate their mobility, self-care, usual activities, pain/discomfort and anxiety/depression developed by Euroqol Research Foundation.
  Each of the 5 dimensions comprising the EQ-5D descriptive system is divided into 5 levels of perceived problems:
  Dimension 1: Mobility Dimension 2: Self-Care Dimension 3: Usual Activities Dimension 4: Pain/Discomfort Dimension 5: Anxiety/Depression
  Level 1: indicating no problem Level 2: indicating slight problems Level 3: indicating moderate problems Level 4: indicating severe problems Level 5: indicating extreme problems
  A total of 3,125 possible health states is defined in this way. Each state is referred to in terms of a 5 digit code.
  Lowest Score: 11111 (No problems on any of the 5 dimensions) Highest Score: 55555 (Extreme problems on all of the 5 dimensions)
Change in Visual Analogue Scale (VAS) | Pre-Op, Peri-Op, 6-weeks, 3-months, 6-months, 12-months, 24-months post-op
  Health Questionnaire: patient's rate their health state on a scale from 0 to 100.
  Score Range: 0-100mm
  Low Score = Lower Pain Intensity High Score = Greater Pain Intensity
Change in Oswestry Disability Index (ODI) | Pre-Op, Peri-Op, 6-weeks, 3-months, 6-months, 12-months, 24-months post-op
  10 Question Health Questionnaire where patient's rate their level of back pain.
  Score Range: 0-100%
  Low Score = Minimal Disability High Score = Severe Disability

CONTACTS AND LOCATIONS:
Overall Officials: Hope Donovan, Principal Investigator — MileStone Research Organization
Locations (3):
- United States (3):
  - Dr. Azmi Nasser, Mesa, Arizona
  - Dr. Daniel Hanson, Maple Grove, Minnesota
  - Dr. Louis Saeger, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jasper GP, Francisco GM, Choi DB, Doberstein CE, Telfeian AE. Clinical Benefits of Ultra- Minimally Invasive Spine Surgery in Awake Obese Patients in an Outpatient Setting : A Retrospective Evaluation of Transforaminal Endoscopic Discectomy with Foraminotomy. JSM Neurosurg Spine. 2014;2(5):1041.
- [Background] Ibrahim R, Gohlke K, Decker O. Endoscopic Electrothermic (ESIJ) Procedure of the Sacroiliac Joint 21-Month Follow up Stud¡es.; 2016.
- [Result] Choi WS, Kim JS, Ryu KS, Hur JW, Seong JH, Cho HJ. Endoscopic Radiofrequency Ablation of the Sacroiliac Joint Complex in the Treatment of Chronic Low Back Pain: A Preliminary Study of Feasibility and Efficacy of a Novel Technique. Biomed Res Int. 2016;2016:2834259. doi: 10.1155/2016/2834259. Epub 2016 Dec 25. PMID 28105414
- [Result] Smith AG, Capobianco R, Cher D, Rudolf L, Sachs D, Gundanna M, Kleiner J, Mody MG, Shamie AN. Open versus minimally invasive sacroiliac joint fusion: a multi-center comparison of perioperative measures and clinical outcomes. Ann Surg Innov Res. 2013 Oct 30;7(1):14. doi: 10.1186/1750-1164-7-14. PMID 24172188
- [Result] Pan Z, Ha Y, Yi S, Cao K. Efficacy of Transforaminal Endoscopic Spine System (TESSYS) Technique in Treating Lumbar Disc Herniation. Med Sci Monit. 2016 Feb 18;22:530-9. doi: 10.12659/msm.894870. PMID 26887645
- [Result] Gibson JN, Cowie JG, Iprenburg M. Transforaminal endoscopic spinal surgery: the future 'gold standard' for discectomy? - A review. Surgeon. 2012 Oct;10(5):290-6. doi: 10.1016/j.surge.2012.05.001. Epub 2012 Jun 15. PMID 22705355
- [Result] Jasper GP, Francisco GM, Telfeian AE. Clinical success of transforaminal endoscopic discectomy with foraminotomy: a retrospective evaluation. Clin Neurol Neurosurg. 2013 Oct;115(10):1961-5. doi: 10.1016/j.clineuro.2013.05.033. Epub 2013 Jul 5. PMID 23835307